CLINICAL TRIAL: NCT01197963
Title: A Surgical Approach to the Management of Type II Diabetes Mellitus in Patients With a BMI Between 25-35 kg/m2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB temporarily halted enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Brad Snyder, Assistant Professor - Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-09-0122
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical treatment (Other): Surgical treatment of one arm of the patient population.
  Interventions: Procedure: Sleeve Gastrectomy and Ileal transposition
- Medically controlled group (Other): Managed by endocrinologists using current medical therapy such as pills, injections and life style medication.
  Interventions: Dietary Supplement: dietary and medical management

INTERVENTIONS:
Procedure: Sleeve Gastrectomy and Ileal transposition — Laparoscopic sleeve gastrectomy with ileal transposition
  Arms: Surgical treatment
Dietary Supplement: dietary and medical management — dietary and medical routine management patients are currently following with an endocrinologist.
  Arms: Medically controlled group

SUMMARY:
The purpose of the study is to determine if by performing surgery we can cure Type II Diabetes.

The surgical procedures:

1. a sleeve gastrectomy, cutting out a portion of the stomach, which provides restriction of caloric intake and rapid gastric emptying.
2. ileal transposition which involves repositioning a 150cm segment of the ileum into the jejunum causing improved glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* age- 21-55 years.
* Body Mass Index between 25-35 kf/m2.
* currently being treated for type 2 diabetes mellitus with oral hypoglycemic, insulin or both for the at least 3 years.
* Documented HbA1c>7.5% for at least 3 months.
* Stable weight for 3 months (+/-)
* Evidence of stable medical treatment for diabetes over the past 12 months.
* Able to provide informed consent -Female subject agrees to participate in accepted birth control methods -

Exclusion Criteria:

* Type I diabetes/juvenile onset
* C-Peptid levels below 1.0 ng/ml
* Previous major upper abdominal surgery

  --Pregnant or plans to become pregnant with in the next 12 months
* Current Malignancy
* Severe pulmonary, cardia, or renal disease
* Eating disorders such as bulimia or binge-eating
* Severe mental health disorders such as schizophrenia and bipolar disorder
* Obesity due to other metabolic disorders
* taking appetite suppressants
* currently abusing illicit drugs,alcohol or using tobacco products
* Unable to provide informed consent
* Unwillingness or unable to comply with study procedures
* any condition that deems them unsuitable for the study in the opinion of the investigators

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Serial Postoperative HgA1c levels | 1 month intervals for 3 months then every 3 months there after
  Effectiveness of the transposition to alleviate hyperglycemia will be measured by following serial post operative HbA1c levels. The change from baseline mearusements will be used to determine the outcome. Type 2 diabetes is considered resolved if there is normalization of fasting glucose(<110 mg/dl) normal HbA1c (<6%) and no need for diabetic medications.

SECONDARY OUTCOMES:
Serial Postoperative Lipid Profiles levels | 1 month for the first 3 months then every 3 months there after
  Lipid profiles will be examined at follow up witha goal of total cholesterol <200 mg/dl, low-density lipoprotein (LDL) levels <100 mg/dl, triglyceride levels <150 mg/dl, and high-density lipoprotein (HDL) levels >40 mg/dl. Patients will be fasting for 8 hours and the serum glucose and GLP-1 level will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Brad E Snyder, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas, Bellaire, Texas, United States